CLINICAL TRIAL: NCT04184713
Title: A Clinical Trial With Nutritional Intervention to Evaluate the Effect of an Specific Oral Nutritional Supplement on the Nutritional Status in Patients With Cancer and Malnutrition
Brief Title: Evaluation of the Effect of an Specific Oral Nutritional Supplement on the Nutritional Status in Cancer and Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Adventia Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HULP 5358
Record Dates: First submitted 2019-09-12; First posted 2019-12-04 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2019-09

CONDITIONS: Malnutrition; Cancer; Nutrition Related Cancer
Keywords: malnutrition; cancer; nutrition; nutritional oral supplement; clinical trial
MeSH Terms: conditions — Malnutrition; Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Nutritional intervention and physical activity recommendations. Consumption of 2 tetra paks/day of a specific oral nutritional supplement
  Interventions: Dietary Supplement: Experimental Group
- Control group (Active Comparator): Nutritional intervention and physical activity recommendations. Consumption of 2 tetra paks/day of a specific oral nutritional supplement
  Interventions: Dietary Supplement: Control Group

INTERVENTIONS:
Dietary Supplement: Experimental Group — Nutritional intervention and physical activity recommendations. Consumption of 2 tetra paks/day of a specific oral nutritional supplement (hypercaloric/hyperproteic with fiber and omega-3 enriched, with L-leucine, betaglucans and medium chain triglycerides) for 8 weeks.
  Arms: Experimental Group
Dietary Supplement: Control Group — Nutritional intervention and physical activity recommendations. Consumption of 2 tetra paks/day of a specific oral nutritional supplement (hypercaloric/hyperproteic with fiber) for 8 weeks.
  Arms: Control group

SUMMARY:
Effect of a specific nutritional oral supplement on the nutritional status of patients with cancer and malnutrition

DETAILED DESCRIPTION:
Multicentric, parallel, randomized, double blind and controlled clinical-nutritional study of 8 weeks of duration and 2 study groups of treatment: Experimental group (experimental nutritional oral supplement); and Control group (control nutritional oral supplement) to evaluate the effect on the nutritional and functional status, the quality of life and body composition of patients with cancer and malnutrition undergoint specficic treatment (chemotherapy, radiotherapy, inmunotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 with a cancer diagnosis (any type).
* Subjects who have initiated during the next mont a treatment with chemo and or radiotherapy with or without surgery.
* Having lost more than 5% of body weight in the last 6 months.
* Adequate cultural level and understanding for the clinical trial.
* Signed informed consent.

Exclusion Criteria:

* Subjects who are participating in other clinical trials.
* Subjects with morbid obesity.
* Subjects who will undergo surgery or who will undergo.
* Subjects with cachexia
* Subjects with infection of a cause other than of the tumor
* Subjects with an infectious process
* Subjects with Diabetes Mellitus treated with insulin and/or not controlled
* Subjects with kidney, heart, respiratory or liver disease.
* Subjects with autoimmune diseases.
* Subjects with mental illness or decrease function cognitive.
* Subjects who consume oral supplements or artificial nutrition and who cannot be withdran at least 1 week before startint the study.
* Patients who have consumed food supplements or fortified foods in omega 3 (arginine or nucleotides) during the previous month.
* Patients who reject oral supplements.
* Pregnant or breastfeeding women.
* Allergic to any component of the formula

Min Age: 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Nutritional status | Change from baseline to day 142
  Subjective Global Assessment (SGA)

SECONDARY OUTCOMES:
Diet quality | Change from baseline to day 142
  72h food registry questionaire
Functional status | Change from baseline to day 142
  Dinamometer
Eastern Cooperative Oncology Group Scale (ECOG) | Change from baseline to day 142
  Eastern Cooperative Oncology Group Scale (ECOG)
Body composition | Change from baseline to day 142
  BIA

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gómez Candela, Msc, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Institute for Health Research IdiPAZ, Madrid, Spain